CLINICAL TRIAL: NCT06012539
Title: A Longitudinal Study of Clinical Nurses Caring for Hospitalized Adults With Covid -19
Brief Title: Nurses Caring for Patients With Covid-19
Status: Completed | Type: Observational
Sponsor: Atlantic Health System (Other)
Responsible Party: Principal Investigator, Mildred Kowalski, PhD, RN, Manager, Nursing Research, Atlantic Health System
Other Study IDs: 1605198-6
Record Dates: First submitted 2023-08-23; First posted 2023-08-25 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Nurse; in Northern New Jersey; Providing Care to Adults With Covid-19
Keywords: nurses, interviews, caring for patients with Covid-19
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Qualitative (interviews) — Interviews were held with participants at three different time points, approximately six months apart. Interviews were taped and analyzed for common themes.

SUMMARY:
The main goal of this study was to understand the perceptions of nurses who cared for patients with Covid-19 at the onset of the pandemic in Northeast USA. Private interviews were held three times with each participant, over the period of 18 months. The interviews were examined for common themes and expressions used by nurses to describe such topics as their professional image, memories, and advise to other nurses.

DETAILED DESCRIPTION:
This study was conducted in a single institution. Forty-one (41) nurses were recruited from various units in the medical center. An effort was made to invite nurses from different clinical units, as well as inexperienced and experienced nurses, and males as well as females. To obtain variety in the participants a randomization list (list of names placed in order by a computer) was used to invite nurses. Participants consented and were aware that they would be interviewed three times. The interviews were recorded for transcription and subsequent analysis.

ELIGIBILITY:
Inclusion Criteria:

* RN employed by facility; cared for adult patients with Covid-19 from March - April 2000, consenting

Exclusion Criteria:

* not employed as an RN; did not care for patients with Covid-19 from March-April 2000 at designated facility, does not agree to consent

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: RNs employed at the participating facility, cared for adult patients with Covid-19 in March-April 2020, consenting, participated in three private interviews (taped) over a period of 18 months.
Sampling Method: Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2020-05-22 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2022-12-27 (Actual)

PRIMARY OUTCOMES:
A longitudinal study of clinical nurses caring for hospitalized adults with Covid -19 | 18 months
  41 nurses were interviewed three times to explore perceptions of caring for patients with Covid-19

CONTACTS AND LOCATIONS:
Locations (1):
- Morristown Medical Center, Morristown, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual data because of the confidentiality of this study. A summary of findings will be disseminated by presentation and/or publications.